CLINICAL TRIAL: NCT01511653
Title: Validation and Comparison of Biomarkers for the Early Detection of Colorectal Adenocarcinoma
Brief Title: Validation of Colon Biomarkers for the Early Detection of Colorectal Adenocarcinoma
Acronym: GLNE010
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Early Detection Research Network (Network)
Responsible Party: Principal Investigator, Dean Brenner, Professor Internal Medicine, University of Michigan
Other Study IDs: GLNE010; NCT01585363 (obsolete NCT alias)
Record Dates: First submitted 2012-01-06; First posted 2012-01-18 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: screening colonoscopy; colon cancer early detection; rectal cancer early detection; colorectal cancer prevention; biomarker validation
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two 10 ml red top (serum) tubes Three 10 ml purple top (EDTA)tubes 25 ml of urine 2 Fecal Immunohistochemical Tests (FIT) Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators are undertaking a multi-center, 13000 subject validation study of several biomarkers for early detection of colon cancer. There are stool based biomarkers and blood based biomarkers being validated in this study. The biomarkers will be compared with colonoscopy and with FIT (fecal immunohistochemistry) tests which are the current standards for colon cancer screening. This is an NCI-early Detection Research Network funded project. The population targeted for this study are those persons undergoing colonoscopy for screening. Prior to colonoscopy or even prepping for colonoscopy, subjects will provide blood and stool samples as well as specific data regarding their GI and general medical history and concomitant medications. If subjects are interested in participating, arrangements will be made to see them. The informed consent process will take place, blood will be obtained, data will be obtained, and the stool kit described and given to the subject to take home. Stool samples will be sent back to the University of Michigan using prepaid mailing labels.

DETAILED DESCRIPTION:
The goal of this trial is to estimate the sensitivity and specificity of stool vimentin methylation, serum galectin-3 ligand, and fecal immunochemical testing for colorectal adenocarcinoma, or 2) screen relevant neoplasms (high-grade dysplasia or adenoma with ≥25% villous histologic features or adenoma measuring ≥1 cm in the greatest dimension or sessile serrated polyps measuring 1 cm or more in diameter) as single markers and in combination. Asymptomatic subjects undergoing a colonoscopic procedure for screening for colorectal cancer are eligible. Patients who have a first or second positive fecal immunochemical test, a positive stool guaiac test or a positive Cologuard test are eligible. Up to 2,500 stool blood or Cologuard positive subjects will be recruited on this protocol. Up to an additional 1,000 subjects who have not had previous FIT tests will be recruited. Subjects with a negative stool blood or Cologuard test are not eligible for enrollment. Subjects will meet with research staff prior to initiation of any colonoscopic preparative procedure. After completing informed consent, they will complete Early Detection Research Network (EDRN) data element forms. Blood and urine will be obtained following EDRN standard operating procedures (SOPs). Subjects will be provided with kits to collect stool samples for fecal immunochemical test (FIT) and processing for stool based biomarkers. The collected samples will be shipped to the Central Laboratory at the University of Michigan or German Cancer Research Center (Deutsches Krebsforschungszentrum, DKFZ), Heidelberg, Germany where the stool will be homogenized, aliquoted, and stored at the Umiversity of Michigan CLASS laboratories . The FIT tests will be sent to the Central Laboratory at the University of Michigan or to DKFZ for quantitative analysis following standard operating procedures provided by Eiken Chemical Company. Data from the screening colonoscopy will be obtained. One year after colonoscopy, subjects will be contacted to determine if they have had a neoplastic colorectal diagnosis or other neoplastic events. Data management and protocol coordination will be performed by the Data Management and Coordinating Center (DMCC) of the EDRN along with the GLNE Prevention Research Base at the University of Michigan and will include a Web-based front end and relational database backend, with biosample tracking (VSIMS). Biosamples will be managed in a high quality repository facility at the University of Michigan.

We will estimate sensitivities and specificities and the corresponding confidence intervals of the stool DNA tests and serum/plasma tests for detection of invasive colorectal neoplasms and for screen relevant neoplasias (Aim 1). We will then test the primary hypothesis to confirm the clinical accuracy of a particular biomarker test or panel (Aim 2). The specific primary hypothesis will be defined prior to data analysis based on state of the art information available at that time about candidate biomarkers and tests. Several specific examples of potential primary hypotheses are given to justify study sample size. Finally, several alternative tests and multi-marker panels will be evaluated. (Aim 3). In secondary analysis, we will (a) provide measures of diagnostic accuracy standardized to the age and gender distribution of US population and (b) assess the effect of subject heterogeneity on the marker performance. A primary objective is to establish an archive of appropriately preserved stool, serum, plasma and DNA human biospecimens to be used by EDRN-approved investigators for future validation and biomarker discovery research (Aim 4).

ELIGIBILITY:
Inclusion Criteria:

* Adults 40*+ undergoing a first time colonoscopy for screening OR
* Positive guaiac-based occult blood or fecal immunochemical test (e.g. FOBT, FIT) in the past 12 months (365 days)
* Willing to sign informed consent
* Able to physically tolerate removal of 50 ml of blood
* Willing to collect 2 stool samples

(*age 60 and up in U.S., 50 and up outside US)

Exclusion Criteria:

* Inability to provide informed consent
* History of Inflammatory Bowel Disease
* Overt rectal bleeding within 1 month (30 days) (including due to suspected hemorrhoids)
* Undergone resection of the colon for any indication
* Subjects with known HIV or chronic viral hepatitis (Hepatitis B and C)
* Subjects with known or suspected HNPCC (Lynch Syndrome) or FAP

  * Any cancer within 5 years of enrollment except any of the following:
  * Squamous cell carcinoma of the skin or Basal cell carcinoma of the skin
  * Carcinoma in situ of the cervix, Stages Ia or Ib invasive squamous cell carcinoma of the cervix treated by surgery only. (Excluded if had pelvic radiation)
  * Stage , 0, I or Ia Grade 1 adenocarcinoma of the endometrium treated with surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 13000 asymptomatic subjects aged 50-80 undergoing routine colonoscopic screening for colorectal cancer from community and major medical center outpatient settings across multiple centers and consortia will be recruited.
Sampling Method: Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2011-10 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Measure the sensitivity of a blood based panel of biomarkers relative to fecal immunochemical testing | 12 weeks from enrollment to completion of colonoscopy
  Test the hypothesis that sensitivity of stool vimentin methylation and/ the blood based panel (serum galectin-3 ligand, CEA, methylated genes BCAT1/IKZF1, Hypomethylated LINE1 from circulating cell free DNA) when combined with fecal immunochemical testing (FIT) will significantly improve the sensitivity of FIT for the detection of colorectal adenocarcinoma, and maintain specificity greater than 0.80.

SECONDARY OUTCOMES:
To measure the specificity of a blood based panel of biomarkers relative to fecal immunochemical testing | 12 weeks from enrollment to completion of colonoscopy
  To test the hypothesis that blood based panel (for example, serum galectin-3 ligand, CEA, methylated genes BCAT1/IKZF1, Hypomethylated LINE1 from circulating cell free DNA), at the same sensitivity of that for fecal immunochemical testing (FIT) for the detection of colorectal adenocarcinoma, has a specificity greater than 0.55 with an anticipated specificity ≥ 0.70.
To measure the sensitivity and specificity of a combined panel of blood and stool based biomarkers for the detection of colorectal cancer | 12 weeks from enrollment to completion of colonoscopy
  To test the hypothesis that stool vimentin methylation, the blood based panel (serum galectin-3 ligand, CEA, methylated genes BCAT1/IKZF1, Hypomethylated LINE1 from circulating cell free DNA), when combined will improve the detection of colorectal adenocarcinoma: at sensitivity ≥0.98 it will have a specificity significantly greater than 0.55.

CONTACTS AND LOCATIONS:
Overall Officials: Dean E Brenner, M.D., Principal Investigator — University of Michigan
Locations (9):
- United States (7):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of North Carolina, Chapel Hill, North Carolina
  - Penn State College of Medicine, Hershey, Pennsylvania
  - M.D. Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington
- University of Calgary-Colon Cancer Screening Centre, Calgary, Alberta, Canada
- German Cancer Research Center (DKFZ), Heidelberg, Germany